CLINICAL TRIAL: NCT00473356
Title: Nutritional Effect of an Amino Acid Mixture on Lean Body Mass (LBM) in Post-bariatric Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F061211001; BJ94
Record Dates: First submitted 2007-05-10; First posted 2007-05-15 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Obesity; Post-gastric Bypass
Keywords: Morbid obesity; Lean body mass; amino acid supplement; laparoscopic gastric bypass
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): to receive amino acid supplement
  Interventions: Dietary Supplement: receive amino acid supplement
- 2 (No Intervention): no amino acid supplement

INTERVENTIONS:
Dietary Supplement: receive amino acid supplement — Receive amino acid supplement
  Arms: 1

SUMMARY:
The Focus of this study is to look at the role of nutrition in maintaining lean body mass post-gastric bypass surgery. The purpose of this study is to test whether LBM is increased in those patients receiving a nutritional supplement of amino acids is enhanced when compared to control patients not receiving the supplement.

DETAILED DESCRIPTION:
You are being asked to participate in a pilot (initial) research study designed to test how effectively a nutritional supplement, Juven, helps people keep lean muscle mass (the amount of muscle tissue in your body) and sustain weight loss after gastric bypass surgery. Abbott laboratories, the manufacturer of Juven, sponsors this research study. Juven is commercially available without prescription in the United States.

If you decide to participate, you will have a DEXA scan to check your lean body mass, an indirect calorimetry (your breath is collected for a period of time and is analyzed) test to check your basal metabolic rate (how much energy your body uses at rest), and a blood test to check your certain hormone made by your intestines (bowel or guts). Each of these tests will be run on you three times. Once, before your gastric bypass surgery, once 2 weeks after your surgery and once two months after your surgery.

If you qualify for the study, you will be randomly (like the flip of a coin) assigned by a computer to receive either Juven twice a day by mouth, or to continue with standard care.

As part of your normal post-operative instructions, you should avoid becoming pregnant for two years after your surgery. Acceptable forms of birth control after gastric bypass include barrier methods (condoms, diaphragm, etc.), Depo-Provera (the shot) and Nuva-Ring (Vaginal ring). The birth control pill is not as reliable after gastric bypass because its absorption is unpredictable. The effects of Juven in pregnant women have not been tested. If you should become pregnant, you should stop taking Juven and notify Dr. Clements or his staff.

ELIGIBILITY:
Inclusion Criteria:

* Each person who has been judged to be an acceptable candidate for laparoscopic gastric bypass (LGB) will be asked to participate in this protocol when they are scheduled for the operation.

Exclusion Criteria:

* Age less than 18
* Pregnant females
* Weight greater than the limit of the DEXA table (Patients over 300 pounds)
* Known allergy to any component fo the amino acid supplement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change in LBM | 2 weeks and 2 months post operatively

SECONDARY OUTCOMES:
Change in fasting serum IGF-1, Leptin, Ghrelin, Gastric Inhibitory Polypeptide (GIP), Glucagon-Like Peptide-1 (GLP-1), Insulin, C Reactive Protein, IL-6, albumen, pre-albumin and glucose, and RMR | 2 weeks and 2 months post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Ronald H Clements, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Kirklin Clinic, Birmingham, Alabama, United States